CLINICAL TRIAL: NCT02389478
Title: Oropharyngeal Administration of Colostrum to Very Low Birth Weight Infants：Effects on Secretory Immunoglobulin A
Brief Title: Oropharyngeal Administration of Colostrum to Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FNF201421
Record Dates: First submitted 2015-02-08; First posted 2015-03-17 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Infant, Very Low Birth Weight
Keywords: oropharyngeal; breastmilk; colostrum; human milk; premature infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- colostrums (Experimental): Oropharyngeal administration of colostrums, every 4 hours，continue for 7days
  Interventions: Procedure: Oropharyngeal administration of colostrums
- Normal saline (Other): Oropharyngeal administration of Normal saline,every 4 hours，continue for 7days
  Interventions: Procedure: Oropharyngeal administration of Normal saline

INTERVENTIONS:
Procedure: Oropharyngeal administration of colostrums — rubbing drops of colostrum inside a baby's cheeks using a sterile syringe
  Other Names: oral immune therapy
  Arms: colostrums
Procedure: Oropharyngeal administration of Normal saline — rubbing drops of Normal saline inside a baby's cheeks using a sterile syringe
  Arms: Normal saline

SUMMARY:
The purpose of this study is to explore the effects of Oropharyngeal administration of colostrum to very low birth weight infants on sIgA and lactoferrin, in order to explore the protect immune function of colostrum to very low birth weight infants, to improve the utilization of breast milk and reduce infection rates of very low birth weight infants.

DETAILED DESCRIPTION:
The number of very low born weight infants increased every year.they are suffer from many questions.Recent studies have shown that Oropharyngeal administration of colostrum to very low birth weight infants can reduce the time reach full enteral nutrition .But there are no evidence support that it can promote infants' immune response. The hypothesis of the current study is that Oropharyngeal administration of colostrum to very low birth weight infants may increase the secretion of sIgA in urine and saliva.

The current study adopts randomized, double blind, controlled intervention trial, gives Oropharyngeal administration of colostrums to very low birth weight infants in intervention group and Oropharyngeal administration of Normal saline to control group. All indicators in this study are discrete traits, for sIgA、Lactoferrin number in Saliva and urine， number of CRP，time Begin oral feeding，time up to full enteral feeding， Person's chi-square tests were used for comparisons. For Blood culture results，The number of necrotizing enterocolitis (NEC) occurred， the investigators use Chi-square tests for comparisons between two groups. The study expects that Oropharyngeal administration of colostrum to very low birth weight infants can increase the secretion of sIgA in urine and saliva.

ELIGIBILITY:
Inclusion Criteria:

1. Born weight≤1500g
2. transferred to our hospital within 24 hours after birth
3. the mother can provide colostrum
4. parents of the infants agreed to participate in this study

Exclusion Criteria:

1. The infants suffering from life-threatening conditions ,such as severe heart disease,whose survival time are expected <30d
2. The infants suffering from any kinds of disease,which impact they take human milk by mouth.(such as gastrointestinal malformations, NEC, etc.）
3. human milk is contraindicated

   * An infant whose mother :

     * Is infected with the human immunodeficiency virus (HIV)
     * Is taking antiretroviral medications
     * Has untreated active tuberculosis
     * Is infected with human T-cell lymphotropic virus type l or ll
     * Is using or dependent on an illicit drug except if the breastmilk is medically indicated
     * Is taking prescribed cancer chemotherapy agents contraindicated for breastfeeding
     * Is receiving any medications contraindicated in breast feeding
     * Is receiving diagnostic or therapeutic radioactive isotopes or exposure to radioactive materials (for as long as they are radioactive in the milk)
   * An infant diagnosed with galactosemia, a rare genetic metabolic disorder

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in sIgA at 7 days | at baseline（first time baby in hospital） and at 7 days
  in urine and saliva
Change from Baseline in lactoferrin at 7 days | at baseline（first time baby in hospital） and at 7 days
  in urine and saliva
Change from Baseline in sIgA at 21 days | at baseline（first time baby in hospital） and at 21 days
  in urine and saliva
Change from Baseline in lactoferrin at 21 days | at baseline（first time baby in hospital） and at 21 days
  in urine and saliva

SECONDARY OUTCOMES:
The duration from admission to the start of oral feeding | participants will be followed for the duration of hospital stay, an expected average of 3 days
  when the first time participants start bottle feeding by mouth（>5ml/once）
The duration from the start of enteric feeding to full enteric feeding | participants will be followed for the duration of hospital stay, an expected average of 14 days
  when the volume of milk participants take by mouth up to 140ml/kg/day
The number of participants with necrotizing enterocolitis (NEC) | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhang YuXia, doctor, Study Chair — Children Hospital of Fudan University

REFERENCES:
- [Background] Rodriguez NA, Meier PP, Groer MW, Zeller JM. Oropharyngeal administration of colostrum to extremely low birth weight infants: theoretical perspectives. J Perinatol. 2009 Jan;29(1):1-7. doi: 10.1038/jp.2008.130. Epub 2008 Sep 4. PMID 18769379